CLINICAL TRIAL: NCT04560751
Title: TACE Combined With Lenvatinib for Unresectable Hepatocellular Carcinoma：A Multicenter, Single-armed, Prospective, Observational Study (Prolong)
Brief Title: TACE Combined With Lenvatinib for Unresectable Hepatocellular Carcinoma (Prolong)
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Zhejiang Cancer Hospital (Other)
Responsible Party: Principal Investigator, guoliang shao, Vice President of Zhejiang Cancer Hospital, Zhejiang Cancer Hospital
Other Study IDs: Prolong
Record Dates: First submitted 2020-09-10; First posted 2020-09-23 (Actual); Last update posted 2020-09-23 (Actual); Status verified 2020-09

CONDITIONS: Carcinoma, Hepatocellular
Keywords: Transarterial chemoembolization; Lenvatinib; Carcinoma, Hepatocellular
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — lenvatinib

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Lenvatinib and TACE: Patients in Lenvatinib + TACE group will take oral lenvatinib within ten days after TACE.
  Interventions: Drug: Lenvatinib; Procedure: TACE

INTERVENTIONS:
Drug: Lenvatinib — Lenvatinib capsules will be administered orally, once daily (for patients <60kg, lenvatinib 8mg po; for patients ≥60kg, lenvatinib 12mg po)
Procedure: TACE — TACE will be performed as needed.

SUMMARY:
This is a multicenter, prospective, observational study in which subjects will be treated with lenvatinib combined with TACE in un-resectable HCC patients who had not received systematic treatment or TACE treatment in the past.

DETAILED DESCRIPTION:
Only 30% of HCC patients received radical resection. Most of the patients are in the advanced stage and can only receive palliative treatment such as TACE or systemic treatment. Lenvatinib is a multi-target receptor tyrosine kinase inhibitor (TKI), which mainly inhibits vascular endothelial growth factor(VEGF) receptor-1, 2, 3; fibroblast growth factors(FGF) receptor-1, 2, 3, 4; platelet derived growth factor receptor(PDGFR)α; RET and KIT and showed significant anti-tumor effect in REFLECT study. The purpose of this study is to explore the efficacy and safety of Lenvatinib and TACE in unresectable HCC patients.

ELIGIBILITY:
Inclusion Criteria:

1. Ages of ≥ 18 and ≤ 75 years old.
2. Clinically or histopathologically diagnosed as hepatocellular carcinoma (HCC).
3. China stage IIb-IIIb patients, not suitable for surgical resection.
4. The imaging examination within 2 weeks before interventional therapy showed that there was at least one target lesion that could be measured by CT or MRI, and the lesion was suitable for repeated and accurate measurement.
5. Child-Pugh scores ≤7.
6. ECOG：0-1.
7. Intended to be treated with TACE combined with lenvatinib.
8. Good organ and bone marrow function: Blood routine: WBC>4.0×109/L、Hb>80g/L, PLT>75×109/L, NEUT>1.5×10⁹/L. Blood coagulation function: International normalized ratio (INR)<1.2. Hepatic function: serum albumin (ALB)>3.5 g/dl, total bilirubin (TBIL) <1.5 × normal upper limit (ULN) (Eliminate biliary obstruction), alanine aminotransferase (ALT) or aspartate aminotransferase (AST) < 3 × ULN. Renal dysfunction：serum creatinine (SCR) <1.5× ULN.
9. Agreed to join the clinical trial and sign the informed consent form.

Exclusion Criteria:

1. Hepatobiliary cell carcinoma, mixed cell carcinoma and fibrolamellar hepatocellular carcinoma.
2. With invasion of the main portal vein or vena cava.
3. Received interventional therapy such as TACE within 2 years.
4. Received systematic treatment in the past.
5. Uncontrollable ascites, hepatic encephalopathy or esophagogastric variceal bleeding.
6. Patients with hypertension who cannot be reduced to normal range after antihypertensive treatment (systolic blood pressure > 140mmHg, or diastolic blood pressure > 90 mmHg).
7. Suffering from grade II or above myocardial ischemia or myocardial infarction, poorly controlled arrhythmia or myocardial ischemia or myocardial infarction (The QTc interval ≥ 450ms, QTc interval is calculated by Fridericia formula).
8. There is a history of gastrointestinal bleeding or a clear tendency of gastrointestinal bleeding in the past 3 months, such as esophageal varices at risk of bleeding, local active ulcer lesions, fecal occult blood ≥ (+).
9. Pregnant or lactating women. A fertile patient who is unwilling or unable to use effective contraception.
10. Patients with HIV infection.
11. Suspected allergy to research drugs.
12. Other situations which the researchers considered ineligible for participating in the trial.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Unrecestable CNLC stage IIb-IIIb HCC patients
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2020-09-30 (Estimated); Primary Completion 2021-12-31 (Estimated); Study Completion 2022-08-31 (Estimated)

PRIMARY OUTCOMES:
Objective response rate（ORR） | up to 12 months
  The percentage of patients who have best overall response of complete response (CR) or partial response (PR) according to mRECIST.

SECONDARY OUTCOMES:
Intrahepatic ORR and Extrahepatic ORR | up to 12 months
  The percentage of patients who have best overall response of complete response (CR) or partial response (PR) according to mRECIST intrahepatic or extrahepatic, respectively.
Progression-free survival (PFS) | up to 12 months
  The time from the beginning of treatment of TACE to the time of tumor progression or death from any cause (according to mRECIST standard)
Alpha-fetoprotein (AFP) response rate | up to 12 months
  A decrease in AFP of more than 20% in AFP+ patients treated with lenvatinib is defined as an AFP response.AFP response rate defined as the percentage of AFP response patients in all AFP positive patients.
Time to progression（TTP） | up to 12 months
  The time from the beginning of treatment of TACE to the time of tumor progression. (according to mRECIST standard)
Adverse events(AEs) | up to 18 months
  AEs(adverse events) evaluated by the CTC-AE 5.0

CONTACTS AND LOCATIONS:
Overall Officials: Guoliang Shao, Professor, Study Chair — Zhejiang Cancer Hospital

IPD SHARING:
Plan to Share IPD: No